CLINICAL TRIAL: NCT07186153
Title: Effect of Sodium Glucose Co-transporter 2 Inhibitors on Left Atrial Remodeling in Diabetic Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abanoub Fayoumy Shawky, Doctor, Assiut University
Other Study IDs: Effect of SGLT2 on LAS
Record Dates: First submitted 2025-08-14; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: SGLT 2 Inhibitors
Keywords: left atrial remodelling
MeSH Terms: interventions — empagliflozin; dapagliflozin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Sodium Glucose Co-transporter 2 (SGLT2) Inhibitor — evaluate and follow-up left atrial volume, diastolic function by 2D echocardiography and left atrial strain parameters using speckle-tracking echocardiography in patients with type 2 diabetes mellitus (T2DM) after treatment with SGLT2 inhibitors
  Other Names: Empagliflozin; Dapagliflozin

SUMMARY:
To evaluate and follow-up left atrial volume, diastolic function by 2D echocardiography and left atrial strain parameters using speckle-tracking echocardiography in patients with type 2 diabetes mellitus (T2DM) before and after treatment with SGLT2 inhibitors

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is a chronic metabolic disorder that significantly increases cardiovascular morbidity and mortality. Among the earliest manifestations of diabetic heart disease is subclinical cardiac dysfunction, which includes left atrial (LA) remodeling and impaired LA function.

LA remodeling encompasses changes in atrial size, geometry, wall stress, and mechanical function, and serves as an early marker of diastolic dysfunction and elevated left ventricular (LV) filling pressures.

These changes are key contributors to the development of heart failure, particularly heart failure with preserved ejection fraction (HFpEF)[4]and is closely associated with an increased risk of atrial fibrillation (AF).

Conventional echocardiographic parameters often fail to detect early LA dysfunction. Recent advances have highlighted left atrial strain-measured via speckle tracking echocardiography (STE)-as a more sensitive and early marker of LA dysfunction . LA strain assessment, especially during the reservoir, conduit, and contraction phases, provides insights into atrial compliance, stiffness, and overall diastolic function, often preceding structural alterations.

Sodium-Glucose Cotransporter-2 (SGLT2) inhibitors are a class of antihyperglycemic agents that have demonstrated significant cardiovascular benefits in clinical trials. Beyond glycemic control, these agents have been linked to favorable cardiac remodeling, improved diastolic function, and reduced filling pressures. However, their impact on LA function, particularly as assessed by strain parameters, remains underexplored

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed T2DM on antidiabetic medication not including SGLT2 inhibitors.
* HbA1c ≤ 7%.
* Age 40-75 years.
* Sinus rhythm.
* Informed consent obtained

Exclusion Criteria:

* History of atrial fibrillation or flutter.
* Patients treated with SGLT2 inhibitors.
* Severe mitral valve regurgitation or stenosis.
* Previous myocardial infarction.
* Previous percutaneous coronary intervention(PCI) or coronary artery bypass grafting (CABG).
* LV Ejection fraction <50% .
* Severe renal impairment (eGFR < 30 mL/min/1.73 m²)
* Uncontrolled hypertension (BP > 160/100 mmHg)
* Inadequate echocardiographic windows or incomplete data

Ages: 40 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults aged 40-75 years with a diagnosis of T2DM on stable antidiabetic therapy not including SGLT2 inhibitors
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
follow-up and evaluation of LA remodeling in patients with type-2 diabetes mellitus ( T2DM) before and after treatment with SGLT2 inhibitors | 6 months follow-up
  The study aims evaluation and follow-up of Left Atrial Strain Parameters assessed by Speckle-Tracking Echocardiography (STE) before and after treatment with SGLT2 inhibitors in patients with type-2 diabetes mellitus at Baseline and 6 months follow-up .
  Left atrial strain will be measured using 2D speckle-tracking echocardiography, including reservoir strain (%), conduit strain (%), and contraction strain (%)

REFERENCES:
- [Background] Rehman SU, Rahman F. Evidence-Based Clinical Review on Cardiovascular Benefits of SGLT2 (Sodium-Glucose Co-Transporter Type 2) Inhibitors in Type 2 Diabetes Mellitus. Cureus. 2020 Aug 11;12(8):e9655. doi: 10.7759/cureus.9655. PMID 32802621
- [Background] Yuda S. Current clinical applications of speckle tracking echocardiography for assessment of left atrial function. J Echocardiogr. 2021 Sep;19(3):129-140. doi: 10.1007/s12574-021-00519-8. Epub 2021 Mar 9. PMID 33687616
- [Background] Swoboda PP, McDiarmid AK, Erhayiem B, Ripley DP, Dobson LE, Garg P, Musa TA, Witte KK, Kearney MT, Barth JH, Ajjan R, Greenwood JP, Plein S. Diabetes Mellitus, Microalbuminuria, and Subclinical Cardiac Disease: Identification and Monitoring of Individuals at Risk of Heart Failure. J Am Heart Assoc. 2017 Jul 17;6(7):e005539. doi: 10.1161/JAHA.117.005539. PMID 28716801
- [Background] Nattel S, Burstein B, Dobrev D. Atrial remodeling and atrial fibrillation: mechanisms and implications. Circ Arrhythm Electrophysiol. 2008 Apr;1(1):62-73. doi: 10.1161/CIRCEP.107.754564. No abstract available. PMID 19808395
- [Background] Tadic M, Cuspidi C. Left atrial function in diabetes: does it help? Acta Diabetol. 2021 Feb;58(2):131-137. doi: 10.1007/s00592-020-01557-x. Epub 2020 Jun 9. PMID 32519220
- [Background] Fan W. Epidemiology in diabetes mellitus and cardiovascular disease. Cardiovasc Endocrinol. 2017 Feb 15;6(1):8-16. doi: 10.1097/XCE.0000000000000116. eCollection 2017 Mar. PMID 31646113